CLINICAL TRIAL: NCT03313856
Title: Effect of Oral Administration of a Herbarium Mixture (Guazuma Ulmifolia and Tecoma Stans) on Metabolic Profile in Type 2 Diabetic Patients
Acronym: GUATECO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Maria Guadalupe Ramos Zavala, Clinical Professor, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2017-09-27; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Two study groups were formed that were randomly assigned with the closed envelope technique to the corresponding group. Group Placebo vs. Guazuma ulmifolia plusTecoma stans
Who Masked: Participant, Investigator
Masking Description: Simple random. It was done with a table of numbers using random selection program Excel 2010.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The patients were randomly assigned to received placebo (calcinaned magnesia), 1 capsule before each meal for a period of 90 days.
  Interventions: Drug: Calcinaned magnesia
- Guazuma ulmifolia plus Tecoma stans (Experimental): The patients were randomly assigned to received the herbarium mixture (GU/TS) , 1 capsule of 400mg, before each meal for a period of 90 days.
  Interventions: Drug: Guazuma Ulmifolia plus Tecoma Stans

INTERVENTIONS:
Drug: Guazuma Ulmifolia plus Tecoma Stans — Guazuma ulmifolia (313.6 mg) -Tecoma stans (86.4 mg) = 400 mg per capsule
  Other Names: GUATECO
  Arms: Guazuma ulmifolia plus Tecoma stans
Drug: Calcinaned magnesia — Calcined magnesia 400 mg per capsule
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the effect of oral administration of herbarium mixture Guazuma ulmifolia (GU) and Tecoma stans (TS) on metabolic profile in type 2 diabetic patients.

DETAILED DESCRIPTION:
A randomized, double blind, placebo controlled, clinical trial was carried out 40 type 2 diabetic patients independently of their basal hypoglycemic treatment. At beginning and at end of the study, BMI, waist circumference, a metabolic profile (fasting glucose, HbA1c, lipids and biosecurity profile), were measured. The patients were randomly assigned to receive the herbarium mixture (GU/TS) 1 g before each meal, or placebo for a period of 90 days. All patients received therapy medical nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Signing of letter of consent under written information.
* Men and women with serum glucose of ≥126 and <400 mg / dl and / or HbA1c ≥6.5% and <10%.
* Age between 30 and 60 years.
* BMI between 25 - 39.9 kg / m2.
* With or without pharmacological treatment with oral hypoglycemic agents or insulin
* Stable body weight during the last 3 months (± 5%).
* Women in the follicular phase of the menstrual cycle (days 3 to 8 of the cycle) at the time of the laboratory tests
* Women who do not expect to be pregnant within the next 3 months.

Exclusion Criteria:

* Physical or mental incapacity that makes it impossible to carry out the intervention.
* Uncontrolled thyroid disease
* Women with suspicion or confirmation of pregnancy.
* Women who are breastfeeding.
* Hepatic disease or elevation to double the upper normal value of TGO and TGP.
* Diagnosis of renal insufficiency or creatinine> 1.5 mg / dL or glomerular filtration rate <60 mL / min).
* Known hypersensitivity to calcined magnesia or Guazuma ulmifolia and / or Tecoma stans.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01-10 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2011-05-31 (Actual)

PRIMARY OUTCOMES:
Modification in fasting glucose in patients with type 2 diabetes after of administration of combination with Guazuma ulmifolia and Tecoma stans | 90 days
  In both groups (intervention and placebo ) of 20 patients each , all patients with type 2 diabetes mellitus, glucose was measured in mg/dL, before and after the administration of the combination guazuma ulmifolia (313.6 mg) and tecoma stans (86.4 mg), one capsule before each food for a period of 90 days. The patient was on a 12-hour fast.
Modification in HbA1c in patients with type 2 diabetes after of administration of combination with Guazuma ulmifolia and Tecoma stans | 90 days
  In both groups (intervention and placebo ) of 20 patients each , all patients with type 2 diabetes mellitus, HbA1c was measured in %, before and after the administration of the combination guazuma ulmifolia (313.6 mg) and tecoma stans (86.4 mg), one capsule before each food for a period of 90 days. The patient was on a 12-hour fast.

SECONDARY OUTCOMES:
Change in lipid profile in patients with type 2 diabetes after of administration of combination with Guazuma ulmifolia and Tecoma stans | 90 days
  In both groups (intervention and placebo ) of 20 patients each , all patients with type 2 diabetes mellitus, lipid profile was measured in mg/dL, before and after the administration of the combination guazuma ulmifolia (313.6 mg) and tecoma stans (86.4 mg), one capsule before each food for a period of 90 days. The patient was on a 12-hour fast.
Modification in insulin in patients with type 2 diabetes after of administration of combination with Guazuma ulmifolia and Tecoma stans | 90 days
  In both groups (intervention and placebo ) of 20 patients each, all patients with type 2 diabetes mellitus, insulin was measured in uU/mL, before and after the administration of the combination guazuma ulmifolia (313.6 mg) and tecoma stans (86.4 mg), one capsule before each food for a period of 90 days. The patient was on a 12-hour fast.
Hepatic safety of administration of guazuma, tecoma through the determination of hepatic profile | 90 days
  The hepatic profile was determined through the serum levels of transaminases in U/L (Glutamic oxalacetic transaminase and Glutamic pyruvic transaminase) after of administration during 90 days of the combination guazuma ulmifolia (313.6 mg) and tecoma stans (86.4 mg). The patient was on a 12-hour fast.
Renal safety of administration of guazuma, tecoma through the determination of serum creatinine | 90 days
  The serum creatinine was measured in mg/dL, before and after of administration during 90 days of the combination guazuma ulmifolia (313.6 mg) and tecoma stans (86.4 mg). The patient was on a 12-hour fast.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaufman RJ. Beta-cell failure, stress, and type 2 diabetes. N Engl J Med. 2011 Nov 17;365(20):1931-3. doi: 10.1056/NEJMcibr1109442. No abstract available. PMID 22087686
- [Background] Saisho Y. beta-cell dysfunction: Its critical role in prevention and management of type 2 diabetes. World J Diabetes. 2015 Feb 15;6(1):109-24. doi: 10.4239/wjd.v6.i1.109. PMID 25685282
- [Background] Andrade-Cetto A, Heinrich M. Mexican plants with hypoglycaemic effect used in the treatment of diabetes. J Ethnopharmacol. 2005 Jul 14;99(3):325-48. doi: 10.1016/j.jep.2005.04.019. PMID 15964161
- [Background] Frei B, Baltisberger M, Sticher O, Heinrich M. Medical ethnobotany of the Zapotecs of the Isthmus-Sierra (Oaxaca, Mexico): documentation and assessment of indigenous uses. J Ethnopharmacol. 1998 Sep;62(2):149-65. doi: 10.1016/s0378-8741(98)00051-8. PMID 9741887
- [Background] Leonti M, Sticher O, Heinrich M. Medicinal plants of the Popoluca, Mexico: organoleptic properties as indigenous selection criteria. J Ethnopharmacol. 2002 Aug;81(3):307-15. doi: 10.1016/s0378-8741(02)00078-8. PMID 12127230
- [Background] Roman-Ramos R, Flores-Saenz JL, Partida-Hernandez G, Lara-Lemus A, Alarcon-Aguilar F. Experimental study of the hypoglycemic effect of some antidiabetic plants. Arch Invest Med (Mex). 1991 Jan-Mar;22(1):87-93. PMID 1819981
- [Background] Alonso-Castro AJ, Salazar-Olivo LA. The anti-diabetic properties of Guazuma ulmifolia Lam are mediated by the stimulation of glucose uptake in normal and diabetic adipocytes without inducing adipogenesis. J Ethnopharmacol. 2008 Jul 23;118(2):252-6. doi: 10.1016/j.jep.2008.04.007. Epub 2008 Apr 12. PMID 18487028
- [Background] Cano JH, Volpato G. Herbal mixtures in the traditional medicine of eastern Cuba. J Ethnopharmacol. 2004 Feb;90(2-3):293-316. doi: 10.1016/j.jep.2003.10.012. PMID 15013195
- [Background] Alarcon-Aguilara FJ, Roman-Ramos R, Perez-Gutierrez S, Aguilar-Contreras A, Contreras-Weber CC, Flores-Saenz JL. Study of the anti-hyperglycemic effect of plants used as antidiabetics. J Ethnopharmacol. 1998 Jun;61(2):101-10. doi: 10.1016/s0378-8741(98)00020-8. PMID 9683340
- [Background] Eddouks M, Bidi A, El Bouhali B, Hajji L, Zeggwagh NA. Antidiabetic plants improving insulin sensitivity. J Pharm Pharmacol. 2014 Sep;66(9):1197-214. doi: 10.1111/jphp.12243. Epub 2014 Apr 15. PMID 24730446
- [Background] Zhang JG, Liu Q, Liu ZL, Li L, Yi LT. Antihyperglycemic activity of Anoectochilus roxburghii polysaccharose in diabetic mice induced by high-fat diet and streptozotocin. J Ethnopharmacol. 2015 Apr 22;164:180-5. doi: 10.1016/j.jep.2015.01.050. Epub 2015 Feb 7. PMID 25660333
- [Background] Tukappa N K A, Londonkar RL, Nayaka HB, Kumar C B S. Cytotoxicity and hepatoprotective attributes of methanolic extract of Rumex vesicarius L. Biol Res. 2015 Mar 25;48(1):19. doi: 10.1186/s40659-015-0009-8. PMID 25857314
- [Background] Wang JJ, Zhao R, Liang JC, Chen Y. The antidiabetic and hepatoprotective effects of magnolol on diabetic rats induced by high-fat diet and streptozotocin. Yao Xue Xue Bao. 2014 Apr;49(4):476-81. PMID 24974464
- [Derived] Pascoe-Gonzalez S, Ramos-Zavala MG, Buenrostro Ahued MA, Hernandez-Gonzalez SO, Cardona-Munoz EG, Garcia-Benavides L, Grover-Paez F. Administration of Herbarium Mixture (Guazuma ulmifolia/Tecoma stans) on Metabolic Profile in Type 2 Diabetes Mellitus Patients: A Randomized, Double-Blind, Placebo-Controlled Trial. J Med Food. 2021 May;24(5):527-532. doi: 10.1089/jmf.2020.0082. Epub 2020 Sep 21. PMID 32955964